CLINICAL TRIAL: NCT05596175
Title: Effectiveness of a Novel Intervention (Super Rehab) in Overweight Patients With Atrial Fibrillation (SuRe AF), a Randomised Controlled Trial.
Brief Title: Super-Rehab: a Novel Approach to Treat Atrial Fibrillation
Acronym: SuRe-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); University of Oxford (Other); Biotronik SE & Co. KG (Industry); RUHX (Official NHS Charity for RUH Bath) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RUH Bath NHS SR AF
Record Dates: First submitted 2022-09-27; First posted 2022-10-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation; Overweight and Obesity
Keywords: Lifestyle risk reduction; Exercise; Behavior modifications; Nutrition therapy; Diet; Cardiovascular disease
MeSH Terms: conditions — Atrial Fibrillation; Overweight; Obesity; Risk Reduction Behavior; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients randomized to Usual Care or Super Rehab plus Usual Care
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind either the participant or care providers to their study arm, however the outcome analysis will be undertaken blinded to study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients will continue Usual Care, which will include having medication optimised for adequate heart-rate control, anti-arrhythmic therapy, and anti-coagulation (for stroke-risk) instituted by their treating Cardiologist if indicated by their CHA₂DS₂-VASc Score. Patients who remain significantly symptomatic despite attempts to optimise medical therapy may be referred for further rhythm management strategies, including cardioversion(s) and/or ablation(s) - as per current standard clinical practice. The Cardiologist will also provide routine, verbal one-off lifestyle advice in line with guidance.
- Super Rehab plus Usual Care (Experimental): 12-month Super Rehab programme involving supervised dietary review sessions, 1-to-1 high-intensity exercise sessions and 3-monthly clinical review of AF risk factors, alongside Usual Care (defined above)
  Interventions: Behavioral: Super Rehab

INTERVENTIONS:
Behavioral: Super Rehab — A 12-month healthcare-delivered lifestyle intervention involving exercise, nutritional support and optimisation of AF-related clinical risk factors.
  Arms: Super Rehab plus Usual Care

SUMMARY:
This study proposes to evaluate the effectiveness of a novel lifestyle intervention (Super Rehab), in addition to standard care, for patients with symptomatic atrial fibrillation (AF) requiring rhythm control strategy who are overweight.

As the main driver behind the selection of a rhythm-control strategy for patients with AF, the primary outcome will be an improvement in AF-related symptoms with Super Rehab versus Usual Care only. Secondary outcomes will include the burden of AF, biochemical and cardiac functional and structural changes, and markers of quality-of-life and health resource use.

DETAILED DESCRIPTION:
In this randomised controlled trial (RCT) the investigators will study the efficacy of a novel lifestyle intervention (Super Rehab), in addition to usual care, for patients with symptomatic atrial fibrillation (AF) where are a rhythm-control strategy is being employed who are overweight. Increasing evidence has shown that AF can respond to robust lifestyle change and aggressive risk factor modification, and in some case can in fact regress.

In the majority of cases, the decision to target a rhythm-control strategy for AF is based on the symptom-burden reported by the patient. This in light of the low volume of evidence suggesting any benefits of rhythm-control strategies over rate-control strategies based on prognostic clinical outcomes.

The modifiable cardiovascular (CV) risk factors that increase both CV risk and the frequency of its various forms of disease also impact the development and progression of AF. In addition, patients with multiple CV risk factors are at enhanced risk of both poorer long-term outcomes and earlier failures of traditional rhythm-control strategies.

This RCT study will involve patients who have described symptomatic AF such that their treating team have elected for a rhythm-control strategy (i.e. a combination of anti-arrhythmic therapy ± a referral for a direct current (DC) cardioversion and/or an ablation) who are also overweight (body mass index [BMI] ≥27kg/m2). The BMI criterion acts as a marker of CV risk that may respond to a lifestyle intervention, which has proved sensitive in other studies.

Participants will be randomised to either Super Rehab and Usual Care or to continue Usual Care only. Super Rehab includes a combination of 1:1 supervised high-intensity exercise, dietary advice sessions and 3-monthly clinical reviews to optimise CV risk factor management. The whole programme lasts 12 months. Participants in both arms will undergo imaging, fitness, clinical tests (including blood tests), and complete questionnaires on four occasions during the study.

The primary outcome of the study will assess the difference in AF symptom burden between the two groups. In addition, the study will assess important secondary outcomes that include change in AF burden (i.e. the amount of time spent in AF), quality-of-life and well-being, biochemical, anthropometric, blood pressure and cardiac functional and structural changes.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18
* Symptomatic AF (paroxysmal or persistent <12-months) with a rhythm control management strategy selected including consideration of referral for a cardioversion or ablation forming part of their planned pathway
* BMI ≥27m/kg2

Exclusion Criteria:

* Prognostic coronary artery disease, defined as left main stem >50% stenosis and/or ≥ moderate disease in ≥3 major epicardial vessels requiring revascularisation.
* Unstable angina
* New York Heart Association class III/IV heart failure or severe left ventricular impairment
* Significant cardiomyopathy (as assessed by Cardiologist, e.g. hypertrophic cardiomyopathy or arrhythmogenic right ventricular cardiomyopathy)
* Severe heart valve disease
* Severe hypertension (BP >180/120mmHg) despite optimising anti-hypertensive therapy
* Uncontrolled arrhythmia or higher degree heart block
* History of aortic dissection
* Recent acute pulmonary embolus, deep vein thrombosis, stroke or transient ischaemic attack (<6 months)
* Severe autonomic or peripheral neuropathy
* Significant acute or chronic renal failure that would preclude contrast use at CT
* Significant pulmonary fibrosis or interstitial lung disease (as assessed by a pulmonary physician)
* Physically unable to participate in high-intensity exercise
* Pregnancy
* Prior AF ablation
* A clinically significant ECG abnormality at the screening visit, which in the opinion of the investigators exposes the subject to risk by enrolling in the trial, including but not limited to: sustained ventricular tachycardia, high-grade atrioventricular block (second-degree Mobitz type II or third-degree heart block), evidence of acute ischemia (ST-segment elevation or depression >1 mm), or other arrhythmias deemed clinically significant by the study cardiologist.
* Participation in another intervention-based research study
* Inability to fully understand the instructions provided during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Symptom burden, as defined by the University of Toronto Atrial Fibrillation Severity Scale (AFSS) | Month 12
  As the primary outcome, an atrial fibrillation-specific measure of symptoms and quality of life will be assessed using the University of Toronto Atrial Fibrillation Severity Scale (AFSS) questionnaire. Scores range from 0 to 35, with higher scores indicating greater AF symptom severity. Differences between groups will be assessed at 12 months, with additional assessments conducted and reported at 6- and 15-month time points.

SECONDARY OUTCOMES:
% burden of AF | Month 12
  Differences between groups of the AF burden - defined as the duration of time spent in atrial fibrillation, as assessed via implantable cardiac monitor (ICM) - will be assessed at 12 months, with additional measurements conducted and reported at 6- and 15-month time points.
Duration and number of AF episodes | Month 12
  Differences between groups in AF duration and frequency will be assessed at 12 months, via implantable cardiac monitor (ICM), with additional measurements conducted and reported at 6- and 15-month time points.
Time to first arrhythmia recurrence | Month 12
  Defined as the time from normal rhythm to the earliest documented date of AF, recorded via implantable cardiac monitor (ICM), following a DCCV or ablation where ICM data was available prior to the intervention.
Anthropometrics - Body weight | 12 months
  Change in weight between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6- and 15-month time points.
Anthropometrics - body mass index | Month 12
  Change in body mass index (BMI) between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6- 15-month time points.
Anthropometrics - abdominal waist circumference | Month 12
  Change in abdominal waist circumference between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6- 15-month time points.
Cardiorespiratory fitness | Month 12
  Differences between groups of the measured maximum rate of oxygen consumption attainable during physical exertion (VO2 peak) will be assessed via cardio pulmonary exercise test (CPET) at 12 months, with additional evaluations conducted and reported at 6- and 15-month time points:
Visceral fat | Month 12
  Differences between groups of the measured visceral fat will be assessed at 12 months (via DEXA body composition scan), with additional evaluations conducted and reported at 6- and 15-month time points.
Cardiac structural and functional assessment with echocardiography | Month 12
  Change in left atrial size and strain between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6- and 15-month time points.
CTCA based changes in left atrial structure | Month 12
  Differences in peri-atrial fat volume and inflammatory signal - assessed by cardiac CT - will be evaluated between groups at 12 months
Blood pressure control | Month 12
  Differences between groups in both systolic and diastolic BP control, using a 7-day home blood pressure diary, will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
Serum lipid levels | Month 12
  Differences between groups in serum lipid levels will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
Glucose control (HbA1c) | Month 12
  Differences between groups in serum HbA1c levels will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
Inflammatory marker (high-sensitivity C-reactive protein) | Month 12
  Differences between groups in serum CRP levels will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
Physical activity | 12 months
  Differences in physical activity between groups, as defined by the implantable cardiac monitor (ICM), will be assessed at 12 months with additional evaluations conducted and reported at 6- and 15-month time points.
European Heart Rhythm Association (EHRA) AF-score | Month 12
  The EHRA AF scale ranges from 1 (no symptoms) to 4 (disabling symptoms). Differences between groups will be assessed at 12 months with additional evaluations conducted and reported at the 6- and 15 month time points.
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire | Month 12
  The AFEQT questionnaire involves responses to a 20-item questionnaire that are scored on a 1 to 7 Likert scale (ranging from 1: "Not at all" to 7: "Extremely"). The four subscales of AFEQT are: Symptoms, Daily activities, Treatment concern and Treatment satisfaction. Overall and subscale scores range from 0 for worst to 100 for best quality of life. Differences between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
EuroQol Group (EuroQol) EQ-5D-5L questionnaire | Month 12
  Patient reported health-related quality-of-life will be recorded using the EuroQol EQ-5D-5L questionnaire. Differences between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6-month and 15-month time points.
Hospital Anxiety and Depression Scale (HADS) | Month 12
  Hospital Anxiety and Depression Scale (HADS) questionnaire. Scores range from 0 to 21 with higher scores reflecting a higher degree of anxiety and/or depression. Differences between groups will be assessed at 12 months, with additional evaluations conducted and reported at the 6- and 15-month time points.
ICEpop CAPability measure for Adults (ICECAP-A) | Month 12
  The ICEpop CAPability measure for Adults (ICECAP-A) will assess holistic capability changes over time as part of a health economic assessment. Scores range from 5 to 20, with higher scores reflecting higher levels of capability. Differences between groups will be assessed at 12 months, with additional evaluations conducted and reported at the 6- and 15-month time points.
Resource-use questionnaire | Month 12
  A study-specific resource-use questionnaire will record health economic parameters including medication burden, primary and secondary care interactions, impact of AF on work status, and smoking status. Differences between groups will be assessed at 12 months, with additional evaluations conducted and reported at 6- and 15-month time points.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khavandi, Principal Investigator — Royal United Hospital NHS Foundation Trust
Locations (1):
- Royal United Hospitals Bath NHS Foundation Trust, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing will be reviewed on an individual basis upon request to the research team.

REFERENCES:
- [Derived] Murphy D, Graby J, Smith T, Peacock O, Abramik J, Antoniades C, Rodrigues JCL, Thompson D, Khavandi A. Effectiveness of a novel intervention (Super Rehab) in overweight patients with atrial fibrillation (SuRe AF): protocol for a randomised controlled trial. BMJ Open. 2025 Sep 14;15(9):e103090. doi: 10.1136/bmjopen-2025-103090. PMID 40953861
- See also: Research team website outlining research goals — http://www.ruh.nhs.uk/SuperRehab